CLINICAL TRIAL: NCT01374360
Title: Paroxysmal Nocturnal Hemoglobinuria (PNH) Registry
Status: Completed | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: M07-001
Record Dates: First submitted 2011-04-15; First posted 2011-06-16 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PNH; Paroxysmal Nocturnal hemoglobinuria; Soliris; Eculizumab; Ravulizumab; Ultomiris
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Receiving Soliris or Ultomiris: PNH patients of any age, including minors, that are receiving Soliris or Ultomiris
- Not receiving Soliris or Ultomiris: PNH patients of any age, including minors, that are not receiving Soliris or Ultomiris

SUMMARY:
This study is a collection of data to evaluate safety and characterize progression of Paroxysmal Nocturnal Hemoglobinuria (PNH).

DETAILED DESCRIPTION:
Collection of data to evaluate safety and characterize progression of Paroxysmal Nocturnal Hemoglobinuria (PNH).

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age, including minors, with a diagnosis of PNH or a detected PNH clone, including patients previously treated with Soliris or Ultomiris and withdrawn from treatment. Patients who are minors must have parent/legal guardian consent and must be willing and able to give assent, if applicable as determined by the Ethics Committees/Institutional Review Boards. Upon attaining adulthood, these patients must be re-consented.
* Ability to comprehend and sign consent to have data entered in the PNH Registry.

Exclusion Criteria:

* Inability or unwillingness to sign informed consent.
* Patients currently enrolled in an interventional clinical trial for treatment of PNH cannot be enrolled in the Registry at the same time.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PNH Patients
Sampling Method: Probability Sample
Enrollment: 6061 (Actual)
Dates: Start 2004-10-29 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Evaluate safety data specific to the use of Soliris and Ultomiris | Ongoing (up to 13 years)
  Primary analyses will assess safety endpoints, including occurrence and time to first event for the following: meningococcal infections, infections with serious outcomes, formation of human anti-drug antibodies (ADA) to Soliris and Ultomiris, malignancy, thrombotic events, pulmonary hypertension, impaired renal function, impaired hepatic function, hemolysis, pregnancies, lactation, infusion reactions, bone marrow transplant, serious adverse events, and mortality.

SECONDARY OUTCOMES:
Collect data to characterize the progression of PNH as well as clinical outcomes, mortality and morbidity in Soliris or Ultomiris and non-Soliris or non- Ultomiris treated patients | Ongoing (up to 13 years)
  Secondary analyses will include descriptions of patient populations, PNH specific treatments, concomitant medications, progression of disease, PNH clone sites, clinical symptoms, and clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Phillipe Gustovic, Study Director — Alexion Pharmaceuticals, Inc.
Locations (1):
- Contact the PNH Registry at Alexion Pharmaceuticals, Inc. for worldwide locations., Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dingli D, Maciejewski JP, Larratt L, Go RS, Hochsmann B, Zu K, Gustovic P, Kulagin AD. Relationship of paroxysmal nocturnal hemoglobinuria (PNH) granulocyte clone size to disease burden and risk of major vascular events in untreated patients: results from the International PNH Registry. Ann Hematol. 2023 Jul;102(7):1637-1644. doi: 10.1007/s00277-023-05269-4. Epub 2023 May 18. PMID 37199789
- [Derived] Hill A, de Latour RP, Kulasekararaj AG, Griffin M, Brodsky RA, Maciejewski JP, Marantz JL, Gustovic P, Schrezenmeier H. Concomitant Immunosuppressive Therapy and Eculizumab Use in Patients with Paroxysmal Nocturnal Hemoglobinuria: An International PNH Registry Analysis. Acta Haematol. 2023;146(1):1-13. doi: 10.1159/000526979. Epub 2022 Sep 15. PMID 36108594
- [Derived] Chou WC, Huang WH, Wang MC, Chang CS, Yeh SP, Chiou TJ, Chen YC, Lin TH, Shen MC; Taiwan PNH study group. Characteristics of Taiwanese patients of PNH in the international PNH registry. Thromb J. 2016 Oct 4;14(Suppl 1):39. doi: 10.1186/s12959-016-0094-0. eCollection 2016. PMID 27766064
- [Derived] Kelly RJ, Hochsmann B, Szer J, Kulasekararaj A, de Guibert S, Roth A, Weitz IC, Armstrong E, Risitano AM, Patriquin CJ, Terriou L, Muus P, Hill A, Turner MP, Schrezenmeier H, Peffault de Latour R. Eculizumab in Pregnant Patients with Paroxysmal Nocturnal Hemoglobinuria. N Engl J Med. 2015 Sep 10;373(11):1032-9. doi: 10.1056/NEJMoa1502950. PMID 26352814
- See also: Registry Summary Overview — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=M07-001&attachmentIdentifier=176aaef6-4514-48c2-9ade-ffaae76d3607&fileName=M07-001_Registry_Summary_Overview_Final_19Nov2025.pdf&versionIdentifier=